CLINICAL TRIAL: NCT06415071
Title: Hypertension Longitudinal Data Platform Linked Electronic Health Records and Public Health Follow-up Database (HYLERP) in Tianjin, China
Brief Title: Hypertension Longitudinal Data Platform in Tianjin
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Collaborators: Tianjin Health Care Big Data Ltd. (Unknown); Tianjin Health Commission (Unknown)
Responsible Party: Principal Investigator, Sun Xin, Professor and director of Chinese Evidence-based Medicine Center, West China Hospital
Other Study IDs: HYLERP
Record Dates: First submitted 2024-05-08; First posted 2024-05-16 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Hypertension
Keywords: Longitudinal data platform; Electronic health records; Public health follow-up database
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with hypertension
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Exposures of interest would be clearly defined according to a specific research question and identified from the database

SUMMARY:
Hypertension is one of the leading causes of death globally, and ranks among the top four risk factors for mortality and DALYs in China. However, large-scale population based longitudinal research data source for hypertension is lacking in China. Thus, we aimed to establish the first and most extensive hypertension database in China using healthcare data from the Tianjin city. This hypertension longitudinal data platformlinked electronic medical records (EMR) system 35 stores healthcare data of 1.17 million hypertension patients, from 43 tertiary hospitals and 39 secondary hospitals, along with a public health follow-up management system. Data on demographics, diagnosis, drug prescription, laboratory test, physical examination, and cost information were collected, the median follow-up time was 4.3 [ interquartile range (IQR): 2.7-5.8] years, and the median number of outpatient visits was 32 (IQR: 15-64) per patient. This database can address research needs including, drug utilization pattern analysis, policy implementation evaluation, digital medical device development, and other real world evidence studies. These researches would provide robust evidence to assist improving patient health outcomes and healthcare system decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension first diagnosed between January 1, 2015 and December 31, 2021
* Aged 18 years or older

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our study population consisted of 1,172,280 patients aged 18 years or older with hypertension diagnosed between January 1, 2015 and December 31, 2021 in database. Hypertension was defined as having at least two outpatient diagnoses or one hospital discharge diagnosis of hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 1172280 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence rate of major adverse cardiovascular events | From index diagnosis to the end of study date (Dec 31, 2021)
  The first occurence of stroke, acute myocardial infarcation and heart failure after index diagnosis. Cardiovasuclar events were determned from the first ICD-10 diagnosis code recorded in the database.
Prevalence of composite adervese events | From index diagnosis to the end of study date (Dec 31, 2021)
  Counts of a composite adervese events after diagnosis including cardiac arrhythmia, gout, hyperkalaemia, hypocalaemia, hypotension, angioedema, fall, syncope, acute kidney injury and fracture. All ICD-10 diagnosis codes of adervese events among patients incurred after the index diagnosis were included to calculated the prevalence of adervese events.
Mortality rate | From index diagnosis to the end of study date (Dec 31, 2021)
  The mortality records on patients were linked to the national mortality register information system, all-cause mortality and cardiovascular mortality were idenitified through death reaseon recoded in the mortality information system.
Prescription patterns of antihypertensive medications | From index prescrition to the end of study date (Dec 31, 2021)
  (1) Prescribing rate of different antihypertensive drug classes; (2) Substiution of generic drugs; (3) Number of drug therapy; (4) Different combination therapies; (4) Index prescription patterns and prevalent prescription patterns.
Medical expenditures | through study completion, an average of 7 year (from Jan 2015 to Dec 31, 2021)
  Medical expenditures per outpatient visit or inpatient admission would be calculated including total expenditures, drug expenditures and non-drug related expenditures for patients undergoing treatment of hypertension, dyslipidemia, diabetes and chronic ischemic heart diesease. All medical expenditures statistcis were based on the cost information recorded in the electronic medical records database.

CONTACTS AND LOCATIONS:
Overall Officials: Xin Sun, Phd, Study Director — West China Second University Hospital
Locations (1):
- The West China Hospital of Sichuan university, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
According to the policy of Tianjin Health Commission, research institutions could apply for data access by submitting a formal study protocol, subjetced to approved by the Tianjin Health Care Big Data Ltd. and the Chinese Evidence -based Medicine Center. Ethical review and research registration are mandatory for all studies.